CLINICAL TRIAL: NCT03315871
Title: Phase II Trial of Combination Immunotherapy in Biochemically Recurrent Prostate Cancer
Brief Title: Combination Immunotherapy in Biochemically Recurrent Prostate Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Principal Investigator, Ravi A. Madan, M.D., Principal Investigator, National Cancer Institute (NCI)
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 180005; 18-C-0005
Record Dates: First submitted 2017-10-18; First posted 2017-10-20 (Actual); Results first posted 2025-06-19 (Actual); Last update posted 2025-06-19 (Actual); Status verified 2025-06

CONDITIONS: Prostate Cancer
Keywords: Antigen direct immunotherapy; PSA; Immunotherapy; Immune Response; Checkpoint Inhibitor
MeSH Terms: conditions — Prostatic Neoplasms | interventions — PROSTVAC; Tomography, X-Ray Computed; Magnetic Resonance Imaging

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- 1/Safety Lead-in Combination Therapy (closed December 2018) (Experimental): Prostvac (rilimogene galvacirepvec/rilimogene glafolivec vaccinia) + CV301+ MSB0011359C (M7824)
  Interventions: Biological: Antigen direct immunotherapy: PROSTVAC-V; Biological: Antigen direct immunotherapy: PROSTVAC-F; Drug: MSB0011359C (M7824); Biological: Antigen direct immunotherapy: CV301; Diagnostic Test: CT scan of chest; Diagnostic Test: CT scan of abdomen/pelvis; Diagnostic Test: MRI; Diagnostic Test: Bone scan
- 2/Biochemical Recurrence: Combination Therapy + Surveillance (closed) (Experimental): Surveillance followed by Prostvac ( rilimogene galvacirepvec/rilimogene glafolivec vaccinia) + CV301 then Prostvac + CV301 + MSB0011359C (M7824)
  Interventions: Biological: Antigen direct immunotherapy: PROSTVAC-V; Biological: Antigen direct immunotherapy: PROSTVAC-F; Drug: MSB0011359C (M7824); Biological: Antigen direct immunotherapy: CV301; Diagnostic Test: CT scan of chest; Diagnostic Test: CT scan of abdomen/pelvis; Diagnostic Test: MRI; Diagnostic Test: PSMA; Diagnostic Test: Bone scan
- 3/Biochemical Recurrence: Combination Antigen Direct Immunotherapy +/- Surveillance (Experimental): Surveillance as needed followed by Prostvac (rilimogene galvacirepvec/rilimogene glafolivec vaccinia) + CV301
  Interventions: Biological: Antigen direct immunotherapy: PROSTVAC-V; Biological: Antigen direct immunotherapy: PROSTVAC-F; Biological: Antigen direct immunotherapy: CV301; Diagnostic Test: CT scan of chest; Diagnostic Test: CT scan of abdomen/pelvis; Diagnostic Test: MRI; Diagnostic Test: PSMA; Diagnostic Test: Bone scan

INTERVENTIONS:
Biological: Antigen direct immunotherapy: PROSTVAC-V — Recombinant vaccinia virus vector antigen direct immunotherapy of the genus Orthopoxvirus. Administered by subcutaneous injection.
  Other Names: rilimogene galvacirepvec/rilimogene glafolivec vaccinia
Biological: Antigen direct immunotherapy: PROSTVAC-F — Recombinant fowlpox virus vector Antigen direct immunotherapy of the genus Avipoxvirus. Administered by subcutaneous injection.
  Other Names: rilimogene galvacirepvec/rilimogene glafolivec fowlpox
Drug: MSB0011359C (M7824) — Fully human bifunctional fusion protein that combines immunoglobulin G1 (IgG1) anti-programmed death-ligand 1 (PD-L1) and Transforming growth factor, beta receptor II (TGFbetaRII) as a monoclonal antibody. Administered via intravenous (IV) infusion over 1 hour.
  Other Names: M7824
  Arms: 1/Safety Lead-in Combination Therapy (closed December 2018); 2/Biochemical Recurrence: Combination Therapy + Surveillance (closed)
Biological: Antigen direct immunotherapy: CV301 — Recombinant vaccinia virus Antigen direct immunotherapy of the genus Avipoxvirus. Administered subcutaneously.
Diagnostic Test: CT scan of chest — Screening, prior to Antigen direct immunotherapy, end of study therapy, then every 6 months as long as participants remain in follow-up. And as clinically indicated after one year.
  Other Names: Computed tomography
Diagnostic Test: CT scan of abdomen/pelvis — Screening, prior to Antigen direct immunotherapy, end of study therapy, then every 6 months as long as participants remain in follow-up. And as clinically indicated after one year.
Diagnostic Test: MRI — Screening, prior to Antigen direct immunotherapy, end of study therapy, then every 6 months as long as participants remain in follow-up. And as clinically indicated after one year.
  Other Names: Magnetic resonance imaging
Diagnostic Test: PSMA — Biochemical recurrence group only. Screening, prior to Antigen direct immunotherapy therapy, end of study therapy, then every 6 months as long as participants remain in follow-up. And as clinically indicated after one year.
  Other Names: prostate-specific membrane antigen positron emission tomography scan
  Arms: 2/Biochemical Recurrence: Combination Therapy + Surveillance (closed); 3/Biochemical Recurrence: Combination Antigen Direct Immunotherapy +/- Surveillance
Diagnostic Test: Bone scan — Screening, prior to Antigen direct immunotherapy, end of study therapy, then every 6 months as long as participants remain in follow-up. And as clinically indicated after one year.

SUMMARY:
Background:

Some people with prostate cancer have a rise in prostate-specific antigen (PSA). This can happen even after treatments like radiation and surgery. Androgen deprivation therapy (ADT) drugs and close monitoring are one standard way to treat this group of people. Another way is to monitor people and their PSA values over time. Researchers want to see if a combination of new drugs can help these people.

Objective:

To see if the combination treatment of PROSTVAC (rilimogene galvacirepvec/rilimogene glafolivec vaccinia), CV301, and MSB0011359C (M7824) can induce an anti-tumor impact in people with biochemically recurrent prostate cancer.

Eligibility:

People ages 18 and older with certain kinds of prostate cancer

Design:

Participants will be screened with

* Medical history
* Physical exam
* Blood and urine tests
* A scan of the neck, chest, abdomen, and pelvis
* A bone scan

A sample of tissue that was already taken will be tested. This will confirm the diagnosis, stage, and disease status.

Some participants will have close monitoring with four monthly PSA checks.

All participants will get two study drugs as shots under the skin. They will get the third drug in a vein. They will get the drugs over at least 7 months. Their vital signs will be checked before they get the drugs and for up to 1 hour after.

Participants will have frequent study visits. They will have physical exams, urine and blood tests, and scans.

Participants will return to the clinic about 4 weeks after they stop taking the study drugs. They will have a medical history, physical exam, and blood tests. They may also have long-term follow-up visits.

DETAILED DESCRIPTION:
Background:

Androgen deprivation therapy (ADT) and surveillance are treatment options for prostate cancer patients with biochemical progression after localized therapy (i.e., biochemically recurrent [BCR] prostate cancer). The primary goal in these patients is to prevent morbidity from their cancer that results from disease progression and metastatic disease on conventional imaging.

ADT can lower the prostate-specific antigen (PSA) in these patients, but because of its substantial side effect profile and ambiguous long-term impact, it is generally deferred by most patients until there is a rapid escalation in their PSA.

Immunotherapy presents an alternative option for these patients that is especially attractive because it is not associated with substantial toxicity. Also, since immunotherapy can have lasting effects after treatment due to a sustained activated immune response, patients will not be required to take these treatments indefinitely to potentially benefit clinically.

Current and previous clinical trials have demonstrated that single agent immunotherapy can impact PSA in patients in this population.

The focus of this study is to determine if combination immunotherapy with Antigen direct immunotherapy antigen directed immunotherapy can initiate an immune response in the first 4 months that is then augmented by an immune checkpoint inhibitor in the following 3 months.

In addition to PSA responses (the primary metric in this population), safety, changes in immune responses, and PSA kinetics will also be evaluated.

Objectives:

Primary Objectives:

Safety Lead-In: To evaluate the safety and tolerability of combination immunotherapy in participants with castration-resistant prostate cancer

Biochemical Recurrence: To determine if the combination immunotherapy can induce a 30% decline in PSA in 28% of participants with biochemically recurrent prostate cancer.

Eligibility Criteria (for biochemical recurrence):

Histologically confirmed adenocarcinoma of the prostate

Participants with negative computed tomography (CT) Scan and Tc-99m Bone Scan

Participants with a PSA over 0.8 ng/ml for participants following radical prostatectomy or for participants following definitive radiation therapy: a rise in PSA of >= 2 ng/mL above the nadir

Participants with a PSA doubling time of 5-15 months

No history of active autoimmune disease or history of organ compromising autoimmune disease

Eastern Cooperative Oncology Group (ECOG) 0-1

Safety lead-in cohort will evaluate 6 participants with castration resistant prostate cancer

Design:

Three-arm, non-randomized study

Accrual goal is a total of 37 evaluable participants (6 in an initial safety cohort, 6 participants who received M7824 (MSB0011359C) as part of the initial investigation and 25 homogenously treated participants without M7824) to evaluate response

Participants from a previous study (NCT02649439) with nearly identical eligibility can serve as a contemporary control for secondary endpoints

Following the safety lead-in, all participants will be enrolled and may undergo a surveillance period during which up to 4 consecutive monthly PSA values will be captured by the labs.

After surveillance period, if applicable, participants will be treated with 2 Antigen direct immunotherapy's concurrently, Prostvac (rilimogene galvacirepvec/rilimogene glafolivec) and CV301, during months 1-4. For months 5-7, MSB0011359C [an anti-programmed Cell Death Ligand 1 (PD-L1) antibody (avelumab) with TGF(Beta)-Trap molecule] will be added to the regimen.

-Effective with amendment v7/29/2021, MSB0011359C (M7824) will no longer be given as part of the treatment combination for the Biochemical Recurrence cohort (Arms 3)

Participants will be monitored for on-treatment and post-treatment PSA, immune and imaging responses.

ELIGIBILITY:
* For Safety Lead-in
* INCLUSION CRITERIA:
* Histopathological documentation of prostate cancer confirmed in either the Laboratory of Pathology at the National Institutes of Health (NIH) Clinical Center, or Walter Reed National Military Medical Center prior to enrollment. If no pathologic specimen is available, participants may enroll with a pathologist's report showing a histologic diagnosis of prostate cancer and a clinical course consistent with the disease.
* Recovery to baseline from acute toxicity related to prior therapy, including surgery and radiation. (28 days removed from last systemic therapy, 14 days removed from last radiation therapy).
* Hepatic function eligibility parameters (within 16 days before starting therapy):

  --Bilirubin less than or equal to upper limit of normal (ULN) (OR in participants with Gilbert's syndrome, a total bilirubin less than or equal to 3.0), aspartate aminotransferase (AST) and alanine aminotransferase (ALT) less than or equal to 1.5 times upper limit of normal.
* Adequate renal function defined by an estimated creatinine clearance > 50 mL/min according to the Cockcroft-Gault formula or by measure of creatinine clearance from 24-hour urine collection.
* No other active malignancies within the past 36 months (with the exception of nonmelanoma skin cancers or carcinoma in situ of the bladder) or life-threatening illnesses.
* Willing to travel to the NIH for follow-up visits.
* 18 years of age or older.
* Able to understand and sign informed consent.
* The effects Prostvac (rilimogene galvacirepvec/rilimogene glafolivec) and CV301 on the developing human fetus are unknown. For this reason, men must agree to use highly effective contraception (that is, methods with a failure rate of less than 1% per year) prior to study entry, for the duration of study therapy and at least four months after the last treatment administration. Should a woman become pregnant or suspect she is pregnant while her partner is participating in this study, she should inform her treating physician immediately.
* Additional Inclusion Criteria Specific to Safety Lead-In Cohort

  * Castrate testosterone level (<50ng/dl or 1.7nmol /L)
  * Progressive disease at study entry defined as one or more of the following criteria occurring in the setting of castrate levels of testosterone:

    * Radiographic progression defined as any new or enlarging bone lesions or growing lymph node disease, consistent with prostate cancer

OR

* For Biochemical Recurrence:
* Prostate-specific antigen (PSA) progression defined by sequence of rising values separated by >1 week (2 separate increasing values over a minimum of 2ng/ml (Prostate Cancer Working Group 2 (PCWG2) PSA eligibility criteria). If participants had been on flutamide, PSA progression is documented 4 weeks or more after withdrawal. For participants on bicalutamide or nilutamide disease progression is documented 6 or more weeks after withdrawal.

  --Participants must agree to continuation of androgen deprivation therapy (ADT) with a gonadotropin-releasing hormone agonist/antagonist or bilateral orchiectomy
* Eastern Cooperative Oncology Group (ECOG) performance status of 0-2 (Karnofsky >80%).
* Hematological eligibility parameters (within 16 days before starting therapy):
* Granulocyte count greater than or equal to 1000/mm^3
* Platelet count greater than or equal to 100 000/mm^3
* Hemoglobin (Hgb) greater than or equal to 9 g/dL
* Prothrombin time (PT) less than or equal to 1.5 x ULN
* Activated partial thromboplastin time (aPTT) less than or equal to 1.5 x ULN

Additional Inclusion Criteria Specific to Biochemical Recurrence Cohort

* Biochemical progression defined as follows:

  * For participants following definitive radiation therapy: a rise in PSA of greater than or equal to 2 ng/mL above the nadir (per Radiation Therapy Oncology Group (RTOG) -American Society for Therapeutic Radiation Oncology (ASTRO) consensus criteria)
  * For participants following radical prostatectomy: rising PSA after surgical procedure (participants must have a PSA greater than or equal to 0.8 ng/mL)
* Participants must have a rising PSA as confirmed by 3 values a minimum of 1 week apart over at least a 1 month period of time.
* Participants must have a PSA doubling time of 5-15 months.
* ECOG performance status of 0-1 (Karnofsky greater than or equal to 80%).
* Negative computed tomography (CT) scan/magnetic resonance imaging (MRI) and bone scan for metastatic prostate cancer.
* Baseline testosterone greater than or equal to 100 ng/dl.
* PSA less than or equal to 30 ng/mL.
* Hematological eligibility parameters (within 16 days before starting therapy):

  * Granulocyte count greater than or equal to 1000/mm3
  * Platelet count greater than or equal to 100 000/mm3
  * Hgb greater than or equal to 10 g/dL

EXCLUSION CRITERIA:

* Immunocompromised status due to:

  * Human immunodeficiency virus (HIV) positivity.
  * Active autoimmune diseases such as Addison's disease, Hashimoto's thyroiditis, systemic lupus erythematosus, Sjogren syndrome, scleroderma, myasthenia gravis, Goodpasture syndrome or active Grave's disease.

    * Participants with a history of autoimmunity that has not required systemic immunosuppressive therapy or does not threaten vital organ function including central nervous system (CNS), heart, lungs, kidneys, skin, and gastrointestinal (GI) tract will be allowed.
    * Participants with diabetes type I, vitiligo, or alopecia are allowed.
  * Other immunodeficiency diseases
  * Splenectomy
* Receipt of any organ transplantation, including allogeneic stem-cell transplantation, but with the exception of transplants that do not require immunosuppression (e.g., corneal transplant, hair transplant).
* Chronic administration (defined as daily or every other day for continued use > 14 days) of systemic corticosteroids within 28 days before the first planned dose of investigational therapy. Use of corticosteroids with minimal systemic absorption (e.g., inhaled steroids, nasal sprays, and topical agents) is allowed.
* Serious intercurrent medical illness that, in the judgment of the investigator, would interfere with participants ability to carry out the treatment program.
* Other medications used for urinary symptoms including 5-alpha reductase inhibitors (finasteride and dutasteride) and alternative medications known to alter PSA (e.g. phytoestrogens and saw palmetto).
* History of prior chemotherapy (chemotherapy allowed for lead-in cohort in castration resistant disease.)
* History of prior immunotherapy within the last 3 years (immunotherapy allowed for lead-in cohort in castration resistant disease.)
* Receipt of an investigational agent within 28 days (or 56 days for an antibody-based therapy) before the first planned dose of study drugs.
* Major surgery within 4 weeks prior to enrollment
* History of allergic reactions attributed to compounds of similar chemical or biologic composition to poxviral Antigen direct immunotherapy's (e.g., vaccinia Antigen direct immunotherapy)
* Previous serious adverse reactions to smallpox vaccination
* History of allergic reactions attributed to monoclonal antibodies (grade 3)
* Known allergy to eggs, egg products, aminoglycoside antibiotics (e.g., gentamicin or tobramycin).
* History of atopic dermatitis or active skin condition (acute, chronic, exfoliative) that disrupts the epidermis
* Unable to avoid close contact or household contact with the following high-risk individuals for three weeks after the Day 1 vaccination: (a) children less than or equal to 3 years of age, (b) pregnant or nursing women, (c) individuals with prior or concurrent extensive eczema or other eczemoid skin disorders, or (d) immunocompromised individuals, such as those with HIV.
* Participants who test positive for hepatitis B virus (HBV) or hepatitis C virus (HCV)
* Clinically significant cardiovascular/cerebrovascular disease as follows: cerebral vascular accident/stroke (< 6 months prior to the first planned dose of study drugs), myocardial infarction (< 6 months prior to the first planned dose of study drugs), unstable angina, congestive heart failure (New York Heart Association Classification Class greater than or equal to II), serious cardiac arrhythmia, or uncontrolled hypertension (systolic blood pressure (SBP)>170/diastolic blood pressure (DBP)>105).
* Participants who have received a red cell transfusion within 2 weeks prior to enrollment.
* Participants unwilling to accept blood products as medically indicated.
* Individual tumor lesion(s) in the liver or chest which are 10 cm or larger.

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2018-03-20 (Actual); Primary Completion 2024-06-04 (Actual); Study Completion 2024-06-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Ravi A Madan, M.D., Principal Investigator — National Cancer Institute (NCI)
Locations (1):
- National Institutes of Health Clinical Center, Bethesda, Maryland, United States

IPD SHARING:
Plan to Share IPD: Yes
All individual participant data (IPD) recorded in the medical record will be shared with intramural investigators upon request. In addition, all large-scale genomic sequencing data will be shared with subscribers to the database of Genotypes and Phenotypes (dbGaP).
Supporting Information: Study Protocol, SAP, ICF
Time Frame: Clinical data available during the study and indefinitely. Genomic data are available once genomic data are uploaded per protocol Genomic Data Sharing (GDS) plan for as long as database is active.
Access Criteria: Clinical data will be made available via subscription to Biomedical Translational Research Information System (BTRIS) and with the permission of the study principal investigator (PI). Genomic data are made available via the database of Genotypes and Phenotypes (dbGaP) through requests to the data custodians.

REFERENCES:
- See also: NIH Clinical Center Detailed Web Page — https://clinicalstudies.info.nih.gov/cgi/detail.cgi?B_2018-C-0005.html

RESULTS

PARTICIPANT FLOW:
Groups:
- 1/ Lead-In Cohort (Closed December 2018)/Arm 1/Combination Therapy [Closed December 2018]: Prostvac (rilimogene galvacirepvec/rilimogene glafolivec vaccinia) + CV301+ MSB0011359C (M7824)
  PROSTVAC-V: Recombinant vaccinia virus vector Antigen direct immunotherapy of the genus Orthopoxvirus. Administered by subcutaneous injection.
  PROSTVAC-F: Recombinant fowlpox virus vector Antigen direct immunotherapy of the genus Avipoxvirus. Administered by subcutaneous injection.
  MSB0011359C (M7824): Fully human bifunctional fusion protein that combines immunoglobulin G1 (IgG1) anti-programmed death-ligand 1 (PD-L1) and Transforming growth factor, beta receptor II (TGFbetaRII) as a monoclonal antibody. Administered via intravenous (IV) infusion over 1 hour.
  CV301: Recombinant vaccinia virus Antigen direct immunotherapy of the genus Avipoxvirus. Administered subcutaneously.
- 2/Biochemical Recurrence Cohort/Arm 1/Combination Therapy [Closed March 2021]: Surveillance followed by Prostvac (rilimogene galvacirepvec/rilimogene glafolivec vaccinia) + CV301 then Prostvac + CV301 + MSB0011359C (M7824)
  PROSTVAC-V: Recombinant vaccinia virus vector Antigen direct immunotherapy of the genus Orthopoxvirus. Administered by subcutaneous injection.
  PROSTVAC-F: Recombinant fowlpox virus vector Antigen direct immunotherapy of the genus Avipoxvirus. Administered by subcutaneous injection.
  MSB0011359C (M7824): Fully human bifunctional fusion protein that combines immunoglobulin G1 (IgG1) anti-programmed death-ligand 1 (PD-L1) and Transforming growth factor, beta receptor II (TGFbetaRII) as a monoclonal antibody. Administered via intravenous (IV) infusion over 1 hour.
  CV301: Recombinant vaccinia virus Antigen direct immunotherapy of the genus Avipoxvirus. Administered subcutaneously.
- 2/Biochemical Recurrence Cohort/Arm2/Combo Therapy (Tx)+/Arm3/Combo Antigen Direct Immunotherapy: Surveillance as needed followed by Prostvac (rilimogene galvacirepvec/rilimogene glafolivec vaccinia) + CV301
  PROSTVAC-V: Recombinant vaccinia virus vector Antigen direct immunotherapy of the genus Orthopoxvirus. Administered by subcutaneous injection.
  PROSTVAC-F: Recombinant fowlpox virus vector Antigen direct immunotherapy of the genus Avipoxvirus. Administered by subcutaneous injection.
  CV301: Recombinant vaccinia virus Antigen direct immunotherapy of the genus Avipoxvirus. Administered subcutaneously.
Period: Safety Lead-In
Arm/Group | 1/ Lead-In Cohort (Closed December 2018)/Arm 1/Combination Therapy [Closed December 2018] | 2/Biochemical Recurrence Cohort/Arm 1/Combination Therapy [Closed March 2021] | 2/Biochemical Recurrence Cohort/Arm2/Combo Therapy (Tx)+/Arm3/Combo Antigen Direct Immunotherapy
Started | 6 | 0 | 0
Completed | 6 | 0 | 0
Not Completed | 0 | 0 | 0
Period: PROSTVAC + CV301 + M7824
Arm/Group | 1/ Lead-In Cohort (Closed December 2018)/Arm 1/Combination Therapy [Closed December 2018] | 2/Biochemical Recurrence Cohort/Arm 1/Combination Therapy [Closed March 2021] | 2/Biochemical Recurrence Cohort/Arm2/Combo Therapy (Tx)+/Arm3/Combo Antigen Direct Immunotherapy
Started | 0 | 8 | 0
Completed | 0 | 2 | 0
Not Completed | 0 | 6 | 0
Not completed — Withdrawal by Subject | 0 | 2 | 0
Not completed — Adverse Event | 0 | 2 | 0
Not completed — Physician Decision | 0 | 1 | 0
Not completed — Participant came off study for intercurrent medical illness. | 0 | 1 | 0
Period: PROSTVAC + CV301
Arm/Group | 1/ Lead-In Cohort (Closed December 2018)/Arm 1/Combination Therapy [Closed December 2018] | 2/Biochemical Recurrence Cohort/Arm 1/Combination Therapy [Closed March 2021] | 2/Biochemical Recurrence Cohort/Arm2/Combo Therapy (Tx)+/Arm3/Combo Antigen Direct Immunotherapy
Started | 0 | 0 | 26
Completed | 0 | 0 | 24
Not Completed | 0 | 0 | 2
Not completed — Progressive disease | 0 | 0 | 1
Not completed — An unrelated lymphoma diagnosis requiring therapy | 0 | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- 2/Biochemical Recurrence Cohort/Arm 1/Combination Therapy [Closed March 2021]: Surveillance as defined by the protocol followed by Prostvac (rilimogene galvacirepvec/rilimogene glafolivec vaccinia) + CV301 then Prostvac + CV301 + MSB0011359C (M7824)
  PROSTVAC-V: Recombinant vaccinia virus vector Antigen direct immunotherapy of the genus Orthopoxvirus. Administered by subcutaneous injection.
  PROSTVAC-F: Recombinant fowlpox virus vector Antigen direct immunotherapy of the genus Avipoxvirus. Administered by subcutaneous injection.
  MSB0011359C (M7824): Fully human bifunctional fusion protein that combines immunoglobulin G1 (IgG1) anti-programmed death-ligand 1 (PD-L1) and Transforming growth factor, beta receptor II (TGFbetaRII) as a monoclonal antibody. Administered via intravenous (IV) infusion over 1 hour.
  CV301: Recombinant vaccinia virus Antigen direct immunotherapy of the genus Avipoxvirus. Administered subcutaneously.
- 2/Biochemical Recurrence Cohort/Arm2/Combo Therapy (Tx)+/Arm3/Combo Antigen Direct Immunotherapy: Surveillance as defined by the protocol followed by Prostvac (rilimogene galvacirepvec/rilimogene glafolivec vaccinia) + CV301
  PROSTVAC-V: Recombinant vaccinia virus vector Antigen direct immunotherapy of the genus Orthopoxvirus. Administered by subcutaneous injection.
  PROSTVAC-F: Recombinant fowlpox virus vector Antigen direct immunotherapy of the genus Avipoxvirus. Administered by subcutaneous injection.
  CV301: Recombinant vaccinia virus Antigen direct immunotherapy of the genus Avipoxvirus. Administered subcutaneously.
- Total: Total of all reporting groups
Arm/Group | 1/ Lead-In Cohort (Closed December 2018)/Arm 1/Combination Therapy [Closed December 2018] | 2/Biochemical Recurrence Cohort/Arm 1/Combination Therapy [Closed March 2021] | 2/Biochemical Recurrence Cohort/Arm2/Combo Therapy (Tx)+/Arm3/Combo Antigen Direct Immunotherapy | Total
Number analyzed (Participants) | 6 | 8 | 26 | 40
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0
  Between 18 and 65 years | 2 | 2 | 7 | 11
  >=65 years | 4 | 6 | 19 | 29
Age, Continuous [Mean (Standard Deviation); unit: years] | 64.5 (5.37) | 74.41 (8.38) | 69.22 (6.61) | 69.55 (7.29)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 0 | 0
  Male | 6 | 8 | 26 | 40
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 2 | 2
  Not Hispanic or Latino | 5 | 8 | 24 | 37
  Unknown or Not Reported | 1 | 0 | 0 | 1
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 1 | 1 | 3 | 5
  White | 5 | 7 | 22 | 34
  More than one race | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 1 | 1
Region of Enrollment [Number; unit: participants]
  United States | 6 | 8 | 26 | 40

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants With a Toxicity
Description: Percentage of participants with a toxicity assessed by the Common Terminology Criteria for Adverse Events (CTCAE v4.0). A serious adverse event is an adverse event or suspected adverse reaction that results in death, a life-threatening adverse drug experience, hospitalization, disruption of the ability to conduct normal life functions, congenital anomaly/birth defect or important medical events that jeopardize the patient or subject and may require medical or surgical intervention to prevent one of the previous outcomes mentioned.
Time Frame: At the end of therapy (7 months)
Measure: Number; unit: Percentage of participants
Groups:
- 2/Biochemical Recurrence Cohort/Arm2/Combo Therapy (Tx)+/Arm3/Combo Antigen Direct Immunotherapy: Surveillance as needed followed by Prostvac (rilimogene galvacirepvec/rilimogene glafolivec vaccinia) + CV301
  PROSTVAC-V: Recombinant vaccinia virus vector vaccine of the genus Orthopoxvirus. Administered by subcutaneous injection.
  PROSTVAC-F: Recombinant fowlpox virus vector vaccine of the genus Avipoxvirus. Administered by subcutaneous injection.
  CV301: Recombinant vaccinia virus vaccine of the genus Avipoxvirus. Administered subcutaneously.
Arm/Group | 1/ Lead-In Cohort (Closed December 2018)/Arm 1/Combination Therapy [Closed December 2018] | 2/Biochemical Recurrence Cohort/Arm 1/Combination Therapy [Closed March 2021] | 2/Biochemical Recurrence Cohort/Arm2/Combo Therapy (Tx)+/Arm3/Combo Antigen Direct Immunotherapy
Number analyzed (Participants) | 6 | 8 | 26
Percentage of participants | 6 | 7 | 24

2. Primary Outcome: Prostate Specific Antigen (PSA) Response
Description: Proportion of evaluable participants who experience at least a 30% decline. PSA is a tumor marker in prostate cancer and elevated in participants with this stage of disease. Declines of 30% can be associated with favorable clinical outcomes.
Time Frame: End of treatment (7 months)
Population: 8/40 participants enrolled were not analyzed because they were not evaluable.
Measure: Number; unit: Proportion of participants
Arm/Group | 1/ Lead-In Cohort (Closed December 2018)/Arm 1/Combination Therapy [Closed December 2018] | 2/Biochemical Recurrence Cohort/Arm 1/Combination Therapy [Closed March 2021] | 2/Biochemical Recurrence Cohort/Arm2/Combo Therapy (Tx)+/Arm3/Combo Antigen Direct Immunotherapy
Number analyzed (Participants) | 6 | 2 | 24
Proportion of participants | 0 | 0 | 0

3. Secondary Outcome: Number of Participants With Related and/or Unrelated Grade 3 and Grade 4 Adverse Events.
Description: Number of participants with related and/or unrelated Grade 3 and Grade 4 adverse events assessed by the Common Terminology Criteria for Adverse Events (CTCAE v4.0). Reporting the grade of adverse events noted in each participant and reporting the fraction with grade 3 and grade 4 adverse events.
Time Frame: 6 weeks
Measure: Count of Participants; unit: Participants
Arm/Group | 1/ Lead-In Cohort (Closed December 2018)/Arm 1/Combination Therapy [Closed December 2018] | 2/Biochemical Recurrence Cohort/Arm 1/Combination Therapy [Closed March 2021] | 2/Biochemical Recurrence Cohort/Arm2/Combo Therapy (Tx)+/Arm3/Combo Antigen Direct Immunotherapy
Number analyzed (Participants) | 6 | 8 | 26
Participants
  Grade 3 Related | 1 | 1 | 0
  Grade 4 Related | 0 | 1 | 0
  Grade 3 Unrelated | 1 | 2 | 3
  Grade 4 Unrelated | 0 | 0 | 0

4. Secondary Outcome: Number of Evaluable Participants With Biochemical Recurrence (BCR) With a 20% Change in PSA Doubling Time
Description: PSA Doubling Time (DT) is the time interval (measured in months) it takes for PSA levels to double. PSA DT was calculated using the Memorial Sloan Kettering online PSA Doubling Time calculator. A long PSA DT suggests more indolent disease based on published data. PSA doubling time has been associated with better clinical outcomes in BCR.
  Note that PSA DT is calculated on a per participant basis and thus will be presented as number of evaluable participants with a change in PSA DT. A change in 20% would be considered meaningful and not due to lab variations. Thus, the data for this outcome is presented as number of evaluable participants experiencing a 20% change in PSA DT.
Time Frame: End of treatment after 7 months
Population: The protocol does not pre-specify to only collect and assess this Outcome Measure in safety 1/Lead-In Cohort. Castration-resistant prostate cancer (CRPC) participants in the safety 1/Lead-In Cohort were evaluated for safety & PSA changes. PSA DT is not a relevant clinical parameter in CRPC disease state, therefore that data was not evaluated for this outcome. Beyond safety CRPC participants will only be evaluated in a descriptive manner, which was done with PSA responses in outcome measure#2.
Measure: Count of Participants; unit: Participants
Arm/Group | 2/Biochemical Recurrence Cohort/Arm 1/Combination Therapy [Closed March 2021] | 2/Biochemical Recurrence Cohort/Arm2/Combo Therapy (Tx)+/Arm3/Combo Antigen Direct Immunotherapy
Number analyzed (Participants) | 8 | 26
Participants
  Participants evaluable for change in PSA Doubling Time | 2 | 23
  Participants with greater than 20% increase in PSA Doubling Time | 1 | 11

5. Other Pre Specified Outcome: Number of Participants With Serious and/or Non-serious Adverse Events Assessed by the Common Terminology Criteria for Adverse Events (CTCAE v4.0)
Description: Here is the number of participants with serious and/or non-serious adverse events assessed by the Common Terminology Criteria for Adverse Events (CTCAE v4.0). A non-serious adverse event is any untoward medical occurrence. A serious adverse event is an adverse event or suspected adverse reaction that results in death, a life-threatening adverse drug experience, hospitalization, disruption of the ability to conduct normal life functions, congenital anomaly/birth defect or important medical events that jeopardize the patient or subject and may require medical or surgical intervention to prevent one of the previous outcomes mentioned.
Time Frame: Adverse Events was monitored/assessed from the first study intervention, Study Day 1 of Cycle 1 through 30 days after the study agent (s) was/were administered, an average of 32 weeks.
Measure: Count of Participants; unit: Participants
Arm/Group | 1/ Lead-In Cohort (Closed December 2018)/Arm 1/Combination Therapy [Closed December 2018] | 2/Biochemical Recurrence Cohort/Arm 1/Combination Therapy [Closed March 2021] | 2/Biochemical Recurrence Cohort/Arm2/Combo Therapy (Tx)+/Arm3/Combo Antigen Direct Immunotherapy
Number analyzed (Participants) | 6 | 8 | 26
Participants | 6 | 7 | 25

ADVERSE EVENTS:
Time Frame: All-Cause Mortality was monitored/assessed for an average of 32 days. Adverse Events was monitored/assessed from the first study intervention, Study Day 1 of Cycle 1 through 30 days after the study agent (s) was/were administered, an average of 32 weeks.
Arm/Group | 1/ Lead-In Cohort (Closed December 2018)/Arm 1/Combination Therapy [Closed December 2018] | 2/Biochemical Recurrence Cohort/Arm 1/Combination Therapy [Closed March 2021] | 2/Biochemical Recurrence Cohort/Arm2/Combo Therapy (Tx)+/Arm3/Combo Antigen Direct Immunotherapy
All-Cause Mortality (participants affected / at risk) | 0/6 | 0/8 | 0/26
Serious Adverse Events (participants affected / at risk) | 1/6 | 3/8 | 2/26
Other Adverse Events (participants affected / at risk) | 6/6 | 7/8 | 25/26
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | 1/ Lead-In Cohort (Closed December 2018)/Arm 1/Combination Therapy [Closed December 2018] (N=6) | 2/Biochemical Recurrence Cohort/Arm 1/Combination Therapy [Closed March 2021] (N=8) | 2/Biochemical Recurrence Cohort/Arm2/Combo Therapy (Tx)+/Arm3/Combo Antigen Direct Immunotherapy (N=26)
Abdominal pain (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
CPK increased (Investigations) | 0 (0) | 1 (2) | 0 (0)
Cardiac disorders - Other, specify: Accelerated Junctional Rhythm (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0)
Diarrhea (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Gastrointestinal disorders - Other, specify: Diverticulitis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Infections and infestations - Other, specify: Covid (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Muscle weakness lower limb (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Myocarditis (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0)
Myositis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (2) | 0 (0)
Neoplasms benign, malignant and unspecified (incl cysts and polyps) - Other, specify: Lymphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1)
Stroke (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | 1/ Lead-In Cohort (Closed December 2018)/Arm 1/Combination Therapy [Closed December 2018] (N=6) | 2/Biochemical Recurrence Cohort/Arm 1/Combination Therapy [Closed March 2021] (N=8) | 2/Biochemical Recurrence Cohort/Arm2/Combo Therapy (Tx)+/Arm3/Combo Antigen Direct Immunotherapy (N=26)
Abdominal pain (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Alanine aminotransferase increased (Investigations) | 0 (0) | 1 (3) | 0 (0)
Alkaline phosphatase increased (Investigations) | 0 (0) | 1 (2) | 0 (0)
Allergic rhinitis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0)
Anemia (Blood and lymphatic system disorders) | 0 (0) | 1 (1) | 0 (0)
Anorexia (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 1 (2)
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Aspartate aminotransferase increased (Investigations) | 0 (0) | 2 (3) | 0 (0)
Back pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Blood and lymphatic system disorders - Other, specify: WBC increased (Blood and lymphatic system disorders) | 0 (0) | 1 (1) | 0 (0)
CPK increased (Investigations) | 0 (0) | 1 (3) | 3 (3)
Cardiac troponin I increased (Investigations) | 0 (0) | 1 (1) | 0 (0)
Chills (General disorders) | 1 (1) | 0 (0) | 0 (0)
Colitis (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Constipation (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Cough (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1) | 0 (0)
Diarrhea (Gastrointestinal disorders) | 1 (1) | 1 (1) | 0 (0)
Dry skin (Skin and subcutaneous tissue disorders) | 2 (2) | 1 (1) | 0 (0)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 2 (2) | 0 (0)
Edema limbs (General disorders) | 0 (0) | 2 (3) | 0 (0)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0)
Eye disorders - Other, specify: Corneal abrasion (Eye disorders) | 0 (0) | 0 (0) | 1 (1)
Eye disorders - Other, specify: Vision Decreased (Eye disorders) | 0 (0) | 0 (0) | 1 (1)
Fall (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
Fatigue (General disorders) | 2 (2) | 3 (4) | 14 (34)
Fever (General disorders) | 1 (1) | 0 (0) | 0 (0)
Flu like symptoms (General disorders) | 3 (5) | 5 (13) | 14 (33)
Headache (Nervous system disorders) | 1 (3) | 0 (0) | 1 (1)
Hematuria (Renal and urinary disorders) | 2 (2) | 2 (3) | 1 (1)
Hemoglobinuria (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0)
Hemorrhoidal hemorrhage (Gastrointestinal disorders) | 1 (1) | 1 (1) | 0 (0)
Hoarseness (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0)
Hot flashes (Vascular disorders) | 0 (0) | 1 (1) | 0 (0)
Hyperkalemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1)
Hyperthyroidism (Endocrine disorders) | 0 (0) | 0 (0) | 1 (1)
Hypoalbuminemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0)
Hypokalemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0)
Hypomagnesemia (Metabolism and nutrition disorders) | 0 (0) | 2 (2) | 0 (0)
Hyponatremia (Metabolism and nutrition disorders) | 0 (0) | 1 (2) | 0 (0)
Hypotension (Vascular disorders) | 1 (1) | 0 (0) | 0 (0)
Injection site reaction (General disorders) | 6 (27) | 7 (23) | 24 (104)
Injury, poisoning and procedural complications - Other, specify: Fingertip (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)
Insomnia (Psychiatric disorders) | 0 (0) | 1 (1) | 0 (0)
Lipase increased (Investigations) | 1 (5) | 3 (6) | 0 (0)
Lung infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Lymphocyte count decreased (Investigations) | 0 (0) | 0 (0) | 2 (4)
Muscle weakness lower limb (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (2) | 0 (0)
Musculoskeletal and connective tissue disorder - Other, specify: Left Knee Meniscus Tear (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Musculoskeletal and connective tissue disorder - Other, specify: Shoulder dislocation (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Musculoskeletal and connective tissue disorder (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) — - Other, specify: Slight headaches and neck stiffness/pain
Myalgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 2 (2)
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1) | 0 (0)
Nausea (Gastrointestinal disorders) | 1 (1) | 1 (1) | 2 (2)
Neoplasms benign, malignant and unspecified (incl cysts and polyps) (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0) — - Other, specify: Keratoacanthoma
Neuralgia (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1)
Non-cardiac chest pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 1 (1)
Oral dysesthesia (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Oral hemorrhage (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Oral pain (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Pain (General disorders) | 4 (4) | 0 (0) | 3 (5)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Platelet count decreased (Investigations) | 0 (0) | 2 (2) | 0 (0)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0)
Presyncope (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Productive cough (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0)
Proteinuria (Renal and urinary disorders) | 0 (0) | 0 (0) | 2 (2)
Pruritus (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 2 (3) | 0 (0) | 1 (2)
Respiratory, thoracic and mediastinal disorders - Other, specify: Consolidation (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0)
Serum amylase increased (Investigations) | 1 (3) | 2 (3) | 0 (0)
Sinus bradycardia (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1)
Skin and subcutaneous tissue disorders - Other, specify: Folliculitis (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Skin and subcutaneous tissue disorders - Other, specify: LE diffuse itchy erythema from waist down (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Skin and subcutaneous tissue disorders - Other, specify: Rash (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Skin hyperpigmentation (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Surgical and medical procedures - Other, specify: Cystoscopy, stent placement (Surgical and medical procedures) | 0 (0) | 0 (0) | 1 (1)
Surgical and medical procedures - Other, specify: L knee arthroplasty (Surgical and medical procedures) | 0 (0) | 0 (0) | 1 (1)
Thromboembolic event (Vascular disorders) | 0 (0) | 1 (1) | 0 (0)
Tooth infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Upper respiratory infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Urinary frequency (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0)
Urinary retention (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1)
Urinary urgency (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1)
Vomiting (Gastrointestinal disorders) | 1 (1) | 1 (1) | 1 (1)
Weight loss (Investigations) | 0 (0) | 1 (1) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2023-05-10): https://cdn.clinicaltrials.gov/large-docs/71/NCT03315871/Prot_SAP_000.pdf
  • Informed Consent Form (2023-05-10): https://cdn.clinicaltrials.gov/large-docs/71/NCT03315871/ICF_001.pdf